CLINICAL TRIAL: NCT03153163
Title: A Phase I Study of Pharmacokinetics and Safety of Trastuzumab Emtansine in Chinese Patients With Logically Advanced Inoperable or Metastatic HER2-Positive Breast Cancer Who Have Received Prior Trastuzumab Based Therapy
Brief Title: Study of the Pharmacokinetics and Safety of Trastuzumab Emtansine in Chinese Participants With Locally Advanced Inoperable or Metastatic HER2+ Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP29920
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Trastuzumab Emtansine (Experimental): Participants with HER2-positive LA/MBC who received prior trastuzumab and taxane therapy will receive trastuzumab emtansine.
  Interventions: Drug: Trastuzumab Emtansine

INTERVENTIONS:
Drug: Trastuzumab Emtansine — Trastuzumab emtansine will be administered by IV infusion at a dose of 3.6 milligrams per kilogram (mg/kg) of body weight, every three weeks (Q3W) until death, disease progression or unmanageable toxicity.
  Other Names: RO5304020

SUMMARY:
This is an open-label Phase I study of single-agent trastuzumab emtansine administered by intravenous (IV) infusion. The study will characterize the pharmacokinetics of trastuzumab emtansine and its relevant analytes and the safety of trastuzumab emtansine in Chinese participants with human epidermal growth factor receptor 2 (HER2)-positive locally advanced/metastatic breast cancer (LA/MBC).

ELIGIBILITY:
Inclusion Criteria:

* Prospective centrally-assessed HER2-positive disease (i.e., immunohistochemistry [IHC] 3 + and/or gene amplified [HER2 to CEP 17 ratio ≥ 2] by in situ hybridization [ISH]) through use of archival paraffin-embedded tumor tissue. Both IHC and ISH assays will be performed; however, only one positive result from either method is required for eligibility
* Tumor tissue block or eight unstained freshly cut slides must be available for central laboratory HER2 testing. Archival tumor samples obtained from primary and/or metastatic sites are acceptable
* For participants with bilateral BC, HER2-positive status must be demonstrated in both locations or in a metastatic site
* Histologically or cytologically confirmed invasive breast cancer (BC): incurable, unresectable, LABC previously treated with multimodality therapy or metastatic breast cancer (MBC)
* Prior treatment for BC in the adjuvant, unresectable, locally advanced, or metastatic setting must include taxane, alone or in combination with another agent, and trastuzumab, alone or in combination with another agent in the adjuvant, unresectable, locally advanced, or metastatic setting
* Documented progression of incurable, unresectable LABC or MBC: Progression must occur during or after most recent treatment for LABC or MBC or within 6 months after completing adjuvant therapy
* Baseline disease that must be evaluable per Response Evaluation Criteria for Solid Tumors Version 1.1 (RECIST v1.1). Participants with CNS-only disease are excluded
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1
* Left ventricular ejection fraction (LVEF) ≥50% by either echocardiogram (ECHO) or multiple-gated acquisition (MUGA)

Exclusion Criteria:

* Prior treatment with trastuzumab emtansine, lapatinib, or capecitabine
* Last dose of prior chemotherapy or trastuzumab within 21 days before the first dose of study treatment
* Hormonal therapy within 7 days before the first dose of study treatment
* Treatment with any other anti-cancer therapy/investigational drug (not defined above) within 21 days prior to randomization, except hormone therapy, which can be given up to 7 days prior to randomization; recovery of treatment-related toxicity consistent with other eligibility criteria before the first dose of treatment
* Radiation therapy within 2 weeks before the first dose of study treatment, and with any related acute toxicity (Grade ≥1)
* Brain metastases that are untreated, symptomatic, progressive, or require therapy, such as radiation or surgery, within 28 days before the first dose of study treatment
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, synchronous or previously diagnosed HER2-positive BC, or cancers with a similar curative outcome as those mentioned above
* Peripheral neuropathy Grade ≥3 per National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) v4.03
* History of exposure to the following cumulative doses of anthracyclines as specified below:

  * Doxorubicin > 500 mg/m^2
  * Epirubucin > 720 mg/m^2
  * Mitoxantrone > 120 mg/m^2 If another anthracycline or more than one anthracycline has been used, then the cumulative dose must not exceed the equivalent of 500 mg/m^2 doxorubicin.
* Cardiopulmonary dysfunction as defined by:

  * Uncontrolled hypertension (persistent systolic blood pressure >150 millimeter of mercury (mmHg) and/or diastolic blood pressure >100 mmHg despite anti-hypertensive therapy)
  * Unstable angina or serious cardiac arrhythmia not controlled by medication
  * Baseline LVEF <50% by either ECHO or MUGA scan
  * History of symptomatic congestive heart failure (Grade ≥3 per NCI CTCAE v4.03 or Class ≥II per New York Heart Association criteria)
  * History of LVEF <40% or symptomatic CHF during prior trastuzumab treatment
  * Myocardial infarction within 6 months before the first dose of study treatment
  * Current dyspnea at rest because of complications of advanced malignancy or any medical need for continuous oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve [AUC] of Trastuzumab Emtansine, Total Trastuzumab, N2'-Deacetyl-N2'-(3-Mercapto-1-Oxopropyl)-Maytansine (DM1), Non-reducible Thioether Linkage (MCC)-DM1 and Lys-MCC-DM1 | Pre-dose, 30 minutes (min), 24, 48, 72/96 hours (hr) post-dose, Day 8, 11, 15, 18 post-dose; Pre-dose, 30 min post-dose Cycle 2 Day 1, Cycle 3 Day 1; Pre-dose Cycle 4 Day 1
  AUC will be evaluated and reported for trastuzumab emtansine and its metabolites.
Maximum Serum Concentration (Cmax) Immediately After Dosing of Trastuzumab Emtansine, Total Trastuzumab, N2'-Deacetyl-N2'-(3-Mercapto-1-Oxopropyl)-Maytansine (DM1), Non-reducible Thioether Linkage (MCC)-DM1 and Lys-MCC-DM1 | Pre-dose, 30 minutes (min), 24, 48, 72/96 hours (hr) post-dose, Day 8, 11, 15, 18 post-dose; Pre-dose, 30 min post-dose Cycle 2 Day 1, Cycle 3 Day 1; Pre-dose Cycle 4 Day 1
  Maximum serum concentration (Cmax) immediately after dosing will be evaluated and reported for trastuzumab emtansine and its metabolites.
Minimum (Trough) Concentration (Cmin) of Trastuzumab Emtansine, Total Trastuzumab, N2'-Deacetyl-N2'-(3-Mercapto-1-Oxopropyl)-Maytansine (DM1), Non-reducible Thioether Linkage (MCC)-DM1 and Lys-MCC-DM1 | Pre-dose, 30 minutes (min), 24, 48, 72/96 hours (hr) post-dose, Day 8, 11, 15, 18 post-dose; Pre-dose, 30 min post-dose Cycle 2 Day 1, Cycle 3 Day 1; Pre-dose Cycle 4 Day 1
  Minimum (Trough) Concentration (Cmin) will be evaluated and reported for trastuzumab emtansine and its metabolites.
Clearance (CL) of Trastuzumab Emtansine, Total Trastuzumab, N2'-Deacetyl-N2'-(3-Mercapto-1-Oxopropyl)-Maytansine (DM1), Non-reducible Thioether Linkage (MCC)-DM1 and Lys-MCC-DM1 | Pre-dose, 30 minutes (min), 24, 48, 72/96 hours (hr) post-dose, Day 8, 11, 15, 18 post-dose; Pre-dose, 30 min post-dose Cycle 2 Day 1, Cycle 3 Day 1; Pre-dose Cycle 4 Day 1
  Clearance (CL) will be evaluated and reported for trastuzumab emtansine and its metabolites.
Volume of Distribution at Steady-State (Vss) of Trastuzumab Emtansine, Total Trastuzumab, N2'-Deacetyl-N2'-(3-Mercapto-1-Oxopropyl)-Maytansine (DM1), Non-reducible Thioether Linkage (MCC)-DM1 and Lys-MCC-DM1 | Pre-dose, 30 minutes (min), 24, 48, 72/96 hours (hr) post-dose, Day 8, 11, 15, 18 post-dose; Pre-dose, 30 min post-dose Cycle 2 Day 1, Cycle 3 Day 1; Pre-dose Cycle 4 Day 1
  Volume of distribution at steady-state (Vss) will be evaluated and reported.
Half-Life (t1/2) of Trastuzumab Emtansine, Total Trastuzumab, N2'-Deacetyl-N2'-(3-Mercapto-1-Oxopropyl)-Maytansine (DM1), Non-reducible Thioether Linkage (MCC)-DM1 and Lys-MCC-DM1 | Pre-dose, 30 minutes (min), 24, 48, 72/96 hours (hr) post-dose, Day 8, 11, 15, 18 post-dose; Pre-dose, 30 min post-dose Cycle 2 Day 1, Cycle 3 Day 1; Pre-dose Cycle 4 Day 1
  Half-life (t1/2) will be evaluated and reported.

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) According to National Cancer Institute Common Terminology Criteria for AEs, Version 4.03 (NCI CTCAE V4.03) | Up to (28-42 days) after the last dose of study drug (57 days)
  An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Fudan University Shanghai Cancer Center; Medical Oncology, Shanghai, China